CLINICAL TRIAL: NCT03358290
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Safety and Efficacy of JTE-051 Administered for 12 Weeks in Subjects With Moderate to Severe Plaque Psoriasis (CLEAR-PS)
Brief Title: Study to Evaluate the Safety and Efficacy of JTE-051 in Subjects With Moderate to Severe Plaque Psoriasis
Acronym: CLEAR-PS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty faced with enrollment in the study
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AE051-G-16-007
Record Dates: First submitted 2017-11-17; First posted 2017-11-30 (Actual); Results first posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Plaque Psoriasis; Skin Diseases
Keywords: JTE-051; Psoriasis
MeSH Terms: conditions — Skin Diseases; Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- JTE-051 Dose 1 (Experimental): One dose of study drug by mouth daily for 12 weeks
  Interventions: Drug: JTE-051
- JTE-051 Dose 2 (Experimental): One dose of study drug by mouth daily for 12 weeks
  Interventions: Drug: JTE-051
- JTE-051 Dose 3 (Experimental): One dose of study drug by mouth daily for 12 weeks
  Interventions: Drug: JTE-051
- JTE-051 Dose 4 (Experimental): One dose of study drug by mouth daily for 12 weeks
  Interventions: Drug: JTE-051
- Placebo (Experimental): One dose of study drug by mouth daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JTE-051 — Active drug tablets containing JTE-051
  Arms: JTE-051 Dose 1; JTE-051 Dose 2; JTE-051 Dose 3; JTE-051 Dose 4
Drug: Placebo — Placebo tablets identical in appearance to the active drug tablets
  Arms: Placebo

SUMMARY:
Study to evaluate the efficacy, safety, tolerability and pharmacokinetics of JTE-051 administered for 12 weeks in subjects with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with moderate to severe plaque psoriasis at least 6 months prior to Visit 1
* Plaque-type psoriasis covering ≥10% of body surface area (BSA) at Visit 1 and Visit 2;
* Psoriasis Area and Severity Index (PASI) score ≥12 at Visit 1 and Visit 2;
* Static Physician's Global Assessment (sPGA) score ≥3 at Visit 1 and Visit 2;
* Body Mass Index (BMI) ≤40 at Visit 1.

Exclusion Criteria:

* Medical history of treatment failure to any systemic agents for plaque psoriasis;
* Presence of erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis or other skin conditions at (e.g., clinically-significant eczema or severe acne) that could interfere with study evaluations at Visit 1;
* Presence or history of any itch due to underlying conditions other than plaque psoriasis which cause or influence pruritus of the skin (e.g., drug induced pruritus, significant other systemic diseases with itch) within 12 months prior to Visit 1;
* History of a clinically-significant infection (e.g., that required oral antimicrobial therapy) within 8 weeks prior to Visit 2;
* History of infections requiring hospitalization or parenteral antibiotic, antiviral, antifungal or antiparasitic therapy within 6 months prior to Visit 2 and no history of recurrent infections or conditions predisposing to chronic infections (e.g., bronchiectasis, chronic osteomyelitis);

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (12):
  - First OC Dermatology, Fountain Valley, California
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - University of South Florida - Hospital, Tampa, Florida
  - Atlanta Dermatology Vein and Research Center LLC, Alpharetta, Georgia
  - Advanced Medical Research, PC, Sandy Springs, Georgia
  - Advanced Clinical Research - Dermatology Center of Canyon County, Nampa, Idaho
  - Clinical Research Advantage, Inc., Evansville, Indiana
  - Kansas City Dermatology P.A., Overland Park, Kansas
  - Forest Hills Dermatology Group, Forest Hills, New York
  - Radiant Research, Inc., Anderson, South Carolina
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Dermatology Treatment and Research Center, Dallas, Texas
- Canada (4):
  - Karma Clinical Trials, St. John's, Newfoundland and Labrador
  - Mediprobe Research Inc., London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - David Gratton's Private Practice, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Written informed consent was obtained prior to performing any study-related procedures. A copy of the informed consent was provided to each subject enrolled in this study. To qualify for the study, subjects were required to satisfy defined criteria.
Pre-assignment Details: Following informed consent signing, screening procedures to confirm eligibility were performed during the Screening Period.
  1. Total screened - 55 subjects
  2. Screen failure - 42 subjects
  3. Randomized - 13 subjects
  4. Safety Population - 13 subjects (All subjects randomized in the study were included in the Safety Population).
  The study was terminated early as per the Sponsor decision.
Groups:
- JTE-051 50 mg: JTE-051 50 mg orally once daily for 12 weeks
- JTE-051 100 mg: JTE-051 100 mg orally once daily for 12 weeks
- JTE-051 150 mg: JTE-051 150 mg orally once daily for 12 weeks
- JTE-051 200 mg: JTE-051 200 mg orally once daily for 12 weeks
- Placebo: Placebo orally once daily for 12 weeks
Period: Overall Study
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Started | 2 | 3 | 3 | 3 | 2
Completed | 2 | 2 | 1 | 1 | 1
Not Completed | 0 | 1 | 2 | 2 | 1
Not completed — Study discontinued by Sponsor | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics results are reported for the Safety Population consisting of the randomized subjects who receive at least one dose of the study drug and have at least one post-randomization safety data: 13 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo | Total
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 2 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 3 | 3 | 2 | 12
  >=65 years | 1 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 2 | 0 | 6
  Male | 1 | 3 | 0 | 1 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 1 | 3 | 3 | 2 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1
  White | 2 | 2 | 2 | 3 | 2 | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 2 | 1 | 1 | 0 | 5
  United States | 1 | 1 | 2 | 2 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving a Minimum 75% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI-75) by End-of-treatment (EOT).
Description: The psoriasis area and severity index (PASI) combines the assessment of the severity of lesions (scaling, redness and plaque thickness) and the area affected into a single score in the range of 0.0 (no disease) to 72.0 (maximal disease). The body is divided into four sections: (1) Head and neck; (2) Upper limbs; (3) Trunk (including axillae and groin); and (4) Lower limbs (including buttocks).
  The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
  The PASI-75 response rate is defined as at least 75 percent (%) reduction in PASI score relative to Baseline.
Time Frame: Up to 12 Weeks
Population: Randomized subjects with available data at EOT (measurement at EOT is the last post-baseline measurement up to Week 12). Of the 13 randomized subjects, 1 subject in the JTE-051 150 mg group did not have any post-baseline data. Therefore, 12 subjects were included in the PASI-75 analysis at EOT.
Measure: Number; unit: % of subjects achieving PASI-75
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2
% of subjects achieving PASI-75 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Percent Change From Baseline in PASI Score
Description: The psoriasis area and severity index (PASI) combines the assessment of the severity of lesions (scaling, redness and plaque thickness) and the area affected into a single score in the range of 0.0 (no disease) to 72.0 (maximal disease). The body is divided into four sections: (1) Head and neck; (2) Upper limbs; (3) Trunk (including axillae and groin); and (4) Lower limbs (including buttocks).
  The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
  Percent change was calculated by taking the Week 12 PASI score and subtracting the baseline PASI, and dividing by the baseline PASI, then multiplying by 100 to get the percent change from baseline.
Time Frame: Week 12
Population: Randomized subjects with available data at Week 12. For the JTE-051 200 mg group, number of participants analyzed is 2 (1 subject completed the study and 1 subject did not complete the study but had available Week 12 data).
Measure: Mean (Standard Deviation); unit: % change in PASI Score
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1
% change in PASI Score | -17.51 (3.120) | -27.69 (2.499) | -33.33 (NA) — Data available only for 1 participant. | -34.09 (33.429) | 0.00 (NA) — Data available only for 1 participant.

3. Secondary Outcome: Proportion of Subjects Achieving PASI-50 (50% Improvement From Baseline in PASI)
Description: The psoriasis area and severity index (PASI) combines the assessment of the severity of lesions (scaling, redness and plaque thickness) and the area affected into a single score in the range of 0.0 (no disease) to 72.0 (maximal disease). The body is divided into four sections: (1) Head and neck; (2) Upper limbs; (3) Trunk (including axillae and groin); and (4) Lower limbs (including buttocks).
  The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
  The PASI-50 response rate is defined as at least 50 percent (%) reduction in PASI score relative to Baseline.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: % of subjects achieving PASI-50
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1
% of subjects achieving PASI-50 | 0 | 0 | 0 | 50 | 0

4. Secondary Outcome: Proportion of Subjects Achieving PASI-90 (90% Improvement From Baseline in PASI)
Description: The psoriasis area and severity index (PASI) combines the assessment of the severity of lesions (scaling, redness and plaque thickness) and the area affected into a single score in the range of 0.0 (no disease) to 72.0 (maximal disease). The body is divided into four sections: (1) Head and neck; (2) Upper limbs; (3) Trunk (including axillae and groin); and (4) Lower limbs (including buttocks).
  The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
  The PASI-90 response rate is defined as at least 90 percent (%) reduction in PASI score relative to Baseline.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: % of subjects achieving PASI-90
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1
% of subjects achieving PASI-90 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Proportion of Subjects Achieving PASI-100 (100% Improvement From Baseline in PASI)
Description: The psoriasis area and severity index (PASI) combines the assessment of the severity of lesions (scaling, redness and plaque thickness) and the area affected into a single score in the range of 0.0 (no disease) to 72.0 (maximal disease). The body is divided into four sections: (1) Head and neck; (2) Upper limbs; (3) Trunk (including axillae and groin); and (4) Lower limbs (including buttocks).
  The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
  The PASI-100 response rate is defined as 100 percent (%) reduction in PASI score relative to Baseline.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: % of subjects achieving PASI-100
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1
% of subjects achieving PASI-100 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Proportion of Subjects Who Achieved Static Physician's Global Assessment (sPGA) Score of 0 or 1
Description: The sPGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the redness, thickness and scaling across all psoriatic lesions. Average redness, thickness and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score is calculated as average of the 3 severity (redness, thickness and scaling) scores and rounded to the nearest whole number score to determine the sPGA score (0=cleared; 1=minimal; 2=mild; 3=moderate; and 4=severe).
  For this outcome measure, a score of 0 means no symptoms of psoriasis and a score of 1 means minimal symptoms of psoriasis.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: % of subjects achieving sPGA 0 or 1
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1
% of subjects achieving sPGA 0 or 1 | 0 | 0 | 0 | 50 | 0

7. Secondary Outcome: Change From Baseline in Static Physician's Global Assessment (sPGA) Score
Description: The sPGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the redness, thickness and scaling across all psoriatic lesions. Average redness, thickness and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score is calculated as average of the 3 severity (redness, thickness and scaling) scores and rounded to the nearest whole number score to determine the sPGA score (0=cleared; 1=minimal; 2=mild; 3=moderate; and 4=severe).
  Change from baseline to Week 12 in sPGA was calculated by taking the Week 12 sPGA and subtracting the baseline sPGA.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1
score on a scale | 0.0 (0.00) | -1.0 (0.00) | 0.0 (NA) — Data available only for 1 participant. | -1.5 (0.71) | 0.0 (NA) — Data available only for 1 participant.

8. Secondary Outcome: Percent Change From Baseline in Psoriasis Body Surface Area (BSA)
Description: The total body surface area (BSA) affected by plaque-type psoriasis was obtained from the percentages of areas affected, including head, trunk, upper limbs and lower limbs. Each reported percentage was multiplied by its respective body region corresponding factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4) and the resulting 4 values were added up to obtain the total psoriasis BSA (Range: 0 to 100).
  BSA (%)=0.1Sh + 0.2Sh+0.3St+0.4Sl, where S=body region surface area with psoriasis: h=head; u=upper limbs; t=trunk; l=lower limbs.
  Percent change from baseline to Week 12 in BSA was calculated by taking the Week 12 BSA and subtracting the baseline BSA, then dividing by the baseline BSA and multiplying by 100.
  A negative change from baseline at Week 12 indicates a reduction in the Psoriasis BSA compared to the baseline.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change in Psoriasis BSA
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1
% change in Psoriasis BSA | 0.00 (0.000) | -20.02 (12.099) | 0.00 (NA) — Data available only for 1 participant. | -0.36 (0.516) | 0.00 (NA) — Data available only for 1 participant.

9. Secondary Outcome: Change From Baseline in the Skindex-16 Overall Score
Description: Skindex-16 questionnaire contains 16 questions related to quality of life in subjects with skin disease. It consists of a short 16-item assessment completed by the subject, with each item rated on a 7-point Likert scale (0=never bothered to 6=always bothered). Each raw score is multiplied by 16.667 to transform all responses to a linear scale from 0 (no effect) to 100 (effect experienced all the time). Responses to the Skindex-16 are categorized into 3 subscales: symptom, emotional & functional; their respective scores are expressed in a linear scale from 0 to 100. Overall scale score is an average of 16 items expressed in a linear scale from 0 to 100.
  Change from baseline to Week 12 in the Skindex-16 Overall Score was calculated by taking the Week 12 Skindex-16 Overall Score and subtracting the baseline Skindex-16 Overall Score.
  A negative change from baseline at Week 12 indicates an improvement in the subject's condition compared to the baseline.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1
score on a scale | -5.75 (15.486) | -14.10 (28.709) | -9.40 (NA) — Data available only for 1 participant. | -20.80 (20.648) | 6.20 (NA) — Data available only for 1 participant.

10. Secondary Outcome: Change From Baseline in the Skindex-16 Symptoms Scale Score
Description: Skindex-16 questionnaire contains 16 questions related to quality of life in subjects with skin disease. It consists of a short 16-item assessment completed by the subject, with each item rated on a 7-point Likert scale (0=never bothered to 6=always bothered). Each raw score is multiplied by 16.667 to transform all responses to a linear scale from 0 (no effect) to 100 (effect experienced all the time). Responses to the Skindex-16 are categorized into 3 subscales: symptom, emotional & functional; their respective scores are expressed in a linear scale from 0 to 100. Symptoms scale score is an average of items 1 to 4 expressed in a linear scale from 0 to 100.
  Change from baseline to Week 12 in the Skindex-16 Symptoms Scale Score was calculated by taking the Week 12 Skindex-16 Symptoms Scale Score and subtracting the baseline Skindex-16 Symptoms Scale Score.
  A negative change from baseline at Week 12 indicates an improvement in the subject's condition compared to the baseline.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1
score on a scale | 8.35 (0.071) | -14.60 (56.003) | -16.60 (NA) — Data available only for 1 participant. | -10.40 (14.708) | 16.60 (NA) — Data available only for 1 participant.

11. Secondary Outcome: Change From Baseline in the Skindex-16 Emotions Scale Score
Description: Skindex-16 questionnaire contains 16 questions related to quality of life in subjects with skin disease. It consists of a short 16-item assessment completed by the subject, with each item rated on a 7-point Likert scale (0=never bothered to 6=always bothered). Each raw score is multiplied by 16.667 to transform all responses to a linear scale from 0 (no effect) to 100 (effect experienced all the time). Responses to the Skindex-16 are categorized into 3 subscales: symptom, emotional & functional; their respective scores are expressed in a linear scale from 0 to 100. Emotions scale score is an average of items 5 to 11 expressed in a linear scale from 0 to 100.
  Change from baseline to Week 12 in the Skindex-16 Emotions Scale Score was calculated by taking the Week 12 Skindex-16 Emotions Scale Score and subtracting the baseline Skindex-16 Emotions Scale Score.
  A negative change from baseline at Week 12 indicates an improvement in the subject's condition compared to the baseline.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1
score on a scale | -9.50 (0.000) | -14.30 (20.223) | -14.30 (NA) — Data available only for 1 participant. | -23.85 (33.729) | -2.40 (NA) — Data available only for 1 participant.

12. Secondary Outcome: Change From Baseline in the Skindex-16 Functioning Scale Score
Description: Skindex-16 questionnaire contains 16 questions related to quality of life in subjects with skin disease. It consists of a short 16-item assessment completed by the subject, with each item rated on a 7-point Likert scale (0=never bothered to 6=always bothered). Each raw score is multiplied by 16.667 to transform responses to a linear scale from 0 (no effect) to 100 (effect experienced all the time). Responses to the Skindex-16 are categorized into 3 subscales: symptom, emotional & functional; their respective scores are expressed in a linear scale from 0 to 100. Functioning scale score is an average of items 12 to 16 expressed in a linear scale from 0 to 100.
  Change from baseline to Week 12 in the Skindex-16 Functioning Scale Score was calculated by taking the Week 12 Skindex-16 Functioning Scale Score and subtracting the baseline Skindex-16 Functioning Scale Score. A negative change from baseline at Week 12 indicates an improvement in the subject's condition compared to the baseline.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1
score on a scale | -11.65 (49.427) | -13.35 (18.880) | 3.40 (NA) — Data available only for 1 participant. | -25.00 (7.071) | 10.00 (NA) — Data available only for 1 participant.

13. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events
Description: Subjects in the Safety Population (13, subjects who were randomly assigned to treatment and who received at least one dose of study drug). The study was terminated early as per the Sponsor decision. All randomized subjects were included in the Safety Population.
Time Frame: Up to 16 Weeks
Population: Subjects in the Safety Population (subjects who were randomly assigned to treatment and who received at least one dose of study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 2
Participants
  Number of subjects with TEAEs | 0 | 2 | 2 | 3 | 0
  Number of subjects with no TEAEs | 2 | 1 | 1 | 0 | 2

14. Secondary Outcome: JTE-051 Trough Plasma Concentrations
Description: Trough plasma concentration is the measured concentration at the end of a dosing interval at steady state (taken directly before next administration). Blood samples were collected at specific timepoints to measure trough plasma concentrations of JTE-051 in the subjects randomized to JTE-051 treatment groups.
Time Frame: Week 12
Population: Subjects randomized to JTE-051 treatment groups with available data at Week 12. For the JTE-051 200 mg group, number of participants analyzed is 2 (1 subject completed the study and 1 subject did not complete the study but had available Week 12 data).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg
Number analyzed (Participants) | 2 | 2 | 1 | 2
ng/mL | 184 (70.7) | 51 (72.1) | 377 (NA) — Data available only for 1 participant. | 203 (286.4)

ADVERSE EVENTS:
Time Frame: Up to 16 Weeks
Description: The Safety Population (subjects who were randomly assigned to treatment and who received at least one dose of study drug) was used for safety analysis.
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/3 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/3 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 2/3 | 2/3 | 3/3 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JTE-051 50 mg (N=2) | JTE-051 100 mg (N=3) | JTE-051 150 mg (N=3) | JTE-051 200 mg (N=3) | Placebo (N=2)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early as per the Sponsor decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications at least 60 days prior to public release. The sponsor will have a review period of 60 days and can embargo communications regarding trial results for an additional period of 60 days from the end of sponsor review period. The sponsor may require removal of any and all confidential information (other than study results) in the communication.

DOCUMENTS (2):
  • Study Protocol (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT03358290/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT03358290/SAP_001.pdf